CLINICAL TRIAL: NCT02594683
Title: A Follow-up Study of a Randomised, Controlled, Study to Investigate the Effects of a New Infant Formula Given in the First 12 Months of Life on Growth and Body Composition up to 5 Years of Age
Brief Title: A Follow-up Study to Investigate the Effects of a New Infant Formula on Growth and Body Composition
Acronym: VenusFU
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other); KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: EBB15GL04185
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stools, saliva and blood (optional)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Key Group of Interest: Exclusively formula fed subjects since 1 month of age
- Other-Fed Group: Mixed feeding of formula and breast milk
- Breastfeeding Group: Exclusively breastfeeding at least until 4 months of age

SUMMARY:
A follow-up study of a randomised, controlled, study to investigate the effects of a new infant formula given in the first 12 months of life on growth and body composition up to 5 years of age

DETAILED DESCRIPTION:
A follow-up study of a randomised, controlled, study to investigate the effects of a new infant formula given in the first 12 months of life on growth and body composition up to 5 years of age. Participants from Venus study will be invited to participate in this follow-up study.

Hypothesis: Significant difference in body mass index (BMI) development for subjects who had received infant formula and follow on formula with scGOS/lcFOS/Nuturis® compared to the control product scGOS/lcFOS and standard formula. No significant difference in growth of subjects who had received infant formula and follow on formula with scGOS/lcFOS/Nuturis® compared to the breast-feeding reference group.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the intervention period of VENUS study until 12 months of age or participation in the VENUS study as breast-fed reference group
* Written informed consent from parent(s) or legally acceptable representatives

Exclusion Criteria:

* Investigator's uncertainty about the willingness or ability of the child and parents to comply with the protocol requirements

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participation in the intervention period of VENUS study until 12 months of age or participation in the VENUS study as breast-fed reference group
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | up to 5 years of age

SECONDARY OUTCOMES:
Sum of skin fold thicknesses (triceps, biceps, suprailiac, subscapular) | up to 5 years of age
Z-scores of Weight-for-age | up to 5 years of age
Z-scores of Weight-for-height | up to 5 years of age
Z-scores of Height-for-age | up to 5 years of age
Z-scores of BMI-for-age | up to 5 years of age
Z-score of Head circumference-for-age | up to 5 years of age
Z-score of Mid-upper-arm-circumference-for-age | up to 5 years of age
Z-score of Skinfold-for-age (subscapular, triceps) | up to 5 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Oon Hoe Teoh, MBBS, Principal Investigator — KK Women's and Children's Hospital; Jian Yi Soh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No